CLINICAL TRIAL: NCT00420901
Title: Effect of Chronic Administration of Sildenafil on Endothelial Function in Men With Diabetes
Brief Title: Effect of Chronic PDE5-Inhibition on Endothelial Function in Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSRRM1999/4
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes
Keywords: function; inhibition
MeSH Terms: conditions — Diabetes Mellitus; Inhibition, Psychological | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
chronic PDE5-Inhibition improves endothelial function in diabetics

DETAILED DESCRIPTION:
Evaluation of endothelial function at baseline and after chronic administration of sildenafil in male subjects with diabetes

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* males

Exclusion Criteria:

* females, nitrate use, PDE5-Inhibitors intolerance

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-01; Study Completion 2000-02

PRIMARY OUTCOMES:
Endothelial function responders - Improvement in endothelial function

SECONDARY OUTCOMES:
Changes in vascular inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: giuseppe rosano, md, Study Director — San Raffaele EUR
Locations (1):
- San Raffaele EUR, Roma, Italy